CLINICAL TRIAL: NCT02993549
Title: Multimodality Monitoring Directed Management of Patients Suffering From Traumatic Brain Injury
Brief Title: TBI Multimodal Monitoring Study
Acronym: monTBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adel Helmy, University Lecturer Neurosurgery, University of Cambridge
Other Study IDs: A094233
Record Dates: First submitted 2016-12-07; First posted 2016-12-15 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Traumatic Brain INjury; Microdialysis
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and cerebrospinal fluid if available. Microdialysis samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head injury is a common and devastating condition that can affect people at any stage of their lives. The treatment of severe head injury takes place in intensive care where interventions are designed to protect the brain from further injury and provide the best environment for recovery. A number of different monitors are used after head injury, including a monitor called microdialysis, to measure how the brain is generating energy. Abnormalities in these monitors guide doctors to the right treatments when the brain is at risk of further injury. There are lots of ways that the brain can be injured further after head injury such as raised pressure in the skull from brain swelling, low oxygen levels and low glucose levels. In this study we aim to combine information from all of these monitors to figure out what the underlying problem is and choose the right intervention to treat the problem that is affecting the patient at the time and compare this with previous treatment protocols to see if it improved outcome.

Aim:

To establish and validate a protocol to treat abnormalities in a microdialysis measure called lactate/pyruvate ratio (LPR) that reflects how cells are generating energy, and compare it with patient cohorts not being monitored using the current protocol.

DETAILED DESCRIPTION:
Background:

Traumatic brain injury (TBI, "head injury) is a major cause of morbidity and mortality worldwide (Hyder et al., 2007). During the first four decades of life, trauma is the leading cause of death and TBI is involved in at least half the number of cases (Jennett, 1996). In the UK, 1,500 per 100,000 of the population (total 1 million) attend Accident and Emergency Departments with a head injury per year. Of these, around 135,000 people are admitted each year and there are an estimated 500,000 people (aged 16 - 74) with long term disabilities as a direct result of TBI (Headway, 2016). Approximately 10 per 100,000 per year die from head injury (Jennett and MacMillan, 1981, Hutchinson et al., 1998).

The major determinant of outcome from TBI is the severity of the primary injury, which is irreversible. However, primary injury invariably leads to the activation of cellular and molecular cascades which mediate further secondary injury that evolve over the ensuing hours and days (Masel and DeWitt, 2010) and are therefore amenable to therapeutic intervention. These molecular cascades can lead to brain swelling within the confines of a fixed intracranial compartment, leading to increased intracranial pressure (ICP) and compromising cerebral perfusion pressure (CPP) (Werner and Engelhard, 2007). The control of ICP and maintenance of CPP has been the bedrock of neurointensive care management of TBI for several decades, however, a recent multicenter randomised clinical trial could not show a long-term favorable outcome with ICP guided therapy (Carney et al., 2012).

The Neuro Critical Care Unit (NCCU) in Cambridge is a world leader in TBI monitoring and routinely employs multi-modal monitoring comprising of ICP, brain tissue oxygen and microdialysis monitoring, in every TBI patient. Conceptually, microdialysis monitoring is an attractive method of assessing tissue biochemistry as it provides a direct measure of metabolic substrates at the cellular level at which energy failure occurs. Specifically, the microdialysis derived measure Lactate/Pyruvate Ratio (LPR) is a measure of cellular redox state and therefore the balance between aerobic and anaerobic metabolism. To date, studies in the literature have focused on demonstrating that individual monitoring parameters e.g. microdialysis derived LPR>25 correlate with an unfavorable outcome in multivariate analyses (Sarrafzadeh et al., 2000, Timofeev et al., 2011).

One reason that an ICP monitoring trial has not been proven to deliver improved outcome is that there are several alternative routes to neuronal injury include insufficient oxygen delivery (Nortje and Gupta, 2006), diffusion barrier within tissues (Smielewski et al., 2002), tissue hypoglycaemia (Vespa et al., 2003) and mitochondrial dysfunction (Verweij et al., 2000). Our understanding of these pathophysiological mechanisms has been greatly advanced by the use of multi-modality monitoring including direct measurement of brain tissue oxygen and cerebral microdialysis. In theory, these pathophysiological states could be treated using treatment of ICP lowering therapy, augmenting cerebral perfusion pressure (CPP), increasing oxygen delivery and augmenting glucose delivery. Though, we currently don't know the best way to combine these treatments and they are often used together making independent analysis difficult. Moreover, there is currently no approved therapy for mitochondrial dysfunction, and while some claim that mitochondrial dysfunction is imminent in increased LPR (Nordstrom et al., 2016), the reality is more complex as there will be conditions that are treatable with an increased LPR, but these states need to be better established for clinicians in order to accurately guide treatment (Lazaridis and Robertson, 2016). Previous implementations of guidelines in TBI have shown to improve care and reduce health related cost, something we hope to achieve with our established clinical protocol (Faul et al., 2007).

Overall research design

We propose a treatment algorithm exploring how a standardised clinical protocol that incorporates multi-modality monitoring parameters (intracranial pressure, brain tissue oxygen and microdialysis parameters) can be systematically and rigorously applied in a traumatic brain injury (TBI) patient cohort with deranged brain chemistry (LPR >25).

Our principal outcome metric is the ability for the protocol to improve the LPR, as well as to see how many patients that may be stratified into any of the suggest treatment categories (see below).

Interventions and assessments

Following inclusion, patients will be monitored using the standard clinical monitoring for sedated and ventilated TBI patients which includes an Intracranial Pressure (ICP) monitor device, a brain tissue oxygen monitor (PbO2) and microdialysis to assess brain biochemistry (Le Roux et al., 2014, Hutchinson et al., 2015). While ICP and PbO2 are measured continually, microdialysis samples are measured hourly. If a derangement in LPR is identified (LPR>25), patients will have an increase in monitoring frequency to every 30 minutes. Our primary measure of deranged energy generation at the cellular level is a LPR>25. This threshold has been shown to relate to an unfavourable long-term outcome (Timofeev et al., 2011, Stein et al., 2012). If the LPR>25 on two consecutive samples (to avoid spurious or transient derangements) it will trigger specific treatment strategies depending on the other contemporaneous monitoring modalities. After each intervention, two consecutive microdialysis samples will be taken to confirm whether LPR has been corrected or whether a further step in the protocol needs to be taken. The sequence of interventions has been chosen on the basis of the strength of association of each intervention with LPR in the existing literature (Hutchinson et al., 2015).

STAGE 1: Correction of Intracranial Hypertension; ICP corrected to <20mmHg Raised ICP compromises delivery of both substrate and oxygen to the injured brain, by reducing Cerebral Perfusion Pressure) and is in itself an independent predictor of poor outcome (Marmarou et al., 1991, Bratton et al., 2007b). In the acute setting we will use hypertonic saline (100ml 5% saline by central venous bolus) as a rapid means of reducing ICP (Marko, 2012). This will be followed by an escalation of ICP control measures using our established ICP protocol (Helmy et al., 2007).

STAGE 2: Ensure sufficient Oxygenation; increase PbO2>15mmHg

Increased LPR can reflect ischaemia and in the first instance we will ensure that there is adequate oxygenation by increasing the PbO2>15mmHg. This threshold of PbO2 has been recognised as physiological in the literature (van den Brink et al., 2000). There are two possible limitations to oxygen availability to brain tissue recognised in TBI:

1. Inadequate oxygen delivery (DO2(brain)=Cerebral Blood Flow (CBF) x Oxygen Capacity in Blood) Firstly, we will ensure adequate haemoglobin concentration (>8g/dl) within the blood and normovolemia to ensure adequate oxygen carrying capacity. Cerebral perfusion pressure (CPP) is monitored as a surrogate of CBF and is usually maintained at around 60-80 mmHg using vasopressors in the NCCU. The CPP target will be based on the autoregulatory parameters of the individual patient utilising ICM+ software. The pressure reactivity index (PRx), is a measure of the ability of the cerebral vasculature to autoregulate to differing CPP (Czosnyka et al., 1997). Keeping the patient's CPP in this autoregulatory range has been show in observational studies to improve outcome (Aries et al., 2012, Needham et al., 2016). If the PRx is >0.3, we will increase the CPP by 10-20 mmHg (to a maximum of 80mmHg as per the upper threshold suggested in the BTF guidelines) (Bratton et al., 2007a).
2. Diffusion Barrier Even with adequate oxygen delivery, microcirculatory collapse at the capillary level can lead to tissue hypoxia (Menon et al., 2004). In this circumstance, increasing the partial pressure of oxygen in arterial blood (PaO2) can increase the gradient between oxygen within the blood and the brain tissue and drive oxygen into the tissues (Reinert et al., 2003). This will be achieved by increasing the fractional inspired oxygen (FiO2) by 40% to a maximum FiO2 of 80%.

STAGE 3: Ensure adequate metabolic substrate delivery; increase brain glucose >1.0 mmol/L Glucose is the primary biochemical substrate in order to generate pyruvate through glycolysis. Brain tissue hypoglycaemia, measured using microdialysis, has been shown to be common following TBI, and is correlated with an unfavourable outcome (Stein et al., 2012). If brain tissue glucose levels falls <1.0 mmol/L, we will increase plasma glucose to 7-10 mmol/L, as lower levels have been shown to correlate to brain tissue hypoglacemia (Oddo et al., 2008), using 50% dextrose. Glucose manipulation has previously been demonstrated to improve LPR (Oddo et al., 2008).

STAGE 4: Persistent LPR>25 despite all monitoring modalities normalized; consider mitochondrial dysfunction The mitochondria are the site of oxidative phosphorylation within cells generating Adenine-Tri-Phosphate (ATP) in the presence of oxygen and suitable biochemical substrate (typically pyruvate) in the tricarboxylic acid (TCA) cycle. It has been empirically demonstrated that following TBI, even in the presence of adequate oxygenation and glucose the mitochondria are incapable of utilising these substrates for energy generation(Verweij et al., 2000). In this circumstance, limited amounts of ATP are generated through anaerobic pathways generating lactate as a byproduct, thus increasing the LPR. In this case, LP ratio is increased, but with an a normal pyruvate concentration (>70mmol/l). In this circumstance there are no accepted pharmacological therapies although in the literature both succinate, a component of the tricarboxcylic acid cycle (Ehinger et al., 2016), and Cyclosporin A, a calcineurin inhibitor, (Mbye et al., 2009) have shown potential efficacy against mitochondrial dysfunction, and Cyclosporin A has a proven safety profile in TBI patients (Mazzeo et al., 2009). It will be up to the treating physician to decide if they wish to consider novel neuroprotective agents or metabolic substrates that have shown promising results in the treatment of mitochondrial dysfunction.

Sampling strategies and data collection

Multimodality monitoring parameters are collected in the neuro-critical care unit (NCCU) in real time, including ICP, CPP (PRx) and PbO2 as well as potential treatments provided. Microdialysis parameters, including the brain metabolites glucose, pyruvate, lactate, glycerol and glutamate, will be sampled every 30 minutes by research nurses in the NCCU. When intracranial monitoring is not deemed necessary anymore, it will be discontinued as per conventional management. The number of interventions that the patient receives and any deviation from the protocol will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head injury requiring ICP monitoring
* Age 18-65 years
* Abnormal CT scan

Exclusion Criteria:

* Bilateral fixed and dilated pupils
* Bleeding diathesis
* Thrombocytopenia (platelets < 100)
* Devastating injuries; patient not expected to survive > 24 hours
* Brainstem damage
* Pregnancy
* Involvement in other studies non-observational studies
* MD catheter located in haemorrhagic lesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from traumatic brain injury in need of intracranial monitoring admitted to the neuro-critical care unit at Addenbrooke's hospital, Cambridge, England.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-16 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
LPR <25 | During neuro-critical care (the first 10 days following trauma).
  Decrease of lactate:pyruvate ratio to below 25
Different pathological targets | During the neuro-critical care period (first 10 days after trauma)
  How many patients have the different pathological targets, including 1. Intracranial hypertension (LPR corrected if ICP <20mmHg), 2. Delivery failure (if LPR is corrected when PbO2 is improved and CPP increased). 3.Oxygen Diffusion Barrier (LPR is corrected if PbO2 is increased through FiO2 increase). 4. Neuroglycopenia (LPR is corrected if brain glucose is increased) or 5. Mitochondrial dysfunction (LPR remains increased despite all the therapies applied).

SECONDARY OUTCOMES:
Monitoring correlation | During the neuro-critical care period (first 10 days after trauma)
  Correlation between Microdialysis parameters (glucose (mmol/L), lactate (mmol/L), pyruvate (mmol/L) and glutamate (µmol/L)) and PbO2 (mmHg), ICP (mmHg) and CPP (mmHg)
Functional Outcome | 6 months following injury
  extended Glasgow Outcome Score 6 months following trauma assessed in the outpatient clinic at Addenbrooke's Hospital. Comparison between patients in different pathological targets.
Cytokine concentration in MD | During the neuro-critical care period (first 10 days after trauma)
  Amount of cytokine concentration in microdialysis sample. Comparison between patients in different pathological targets.
Biomarker concentration in serum | During the neuro-critical care (first 10 days after trauma)
  Amount of S100B concentration (µg/L) through serum samples taken twice daily in the neuro-critical care unit. Comparison between patients in different pathological targets.

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital NHS Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Jennett B. Epidemiology of head injury. J Neurol Neurosurg Psychiatry. 1996 Apr;60(4):362-9. doi: 10.1136/jnnp.60.4.362. No abstract available. PMID 8774396
- [Background] Jennett B, MacMillan R. Epidemiology of head injury. Br Med J (Clin Res Ed). 1981 Jan 10;282(6258):101-4. doi: 10.1136/bmj.282.6258.101. PMID 6779889
- [Background] Hutchinson PJ, Kirkpatrick PJ, Addison J, Jackson S, Pickard JD. The management of minor traumatic brain injury. J Accid Emerg Med. 1998 Mar;15(2):84-8. doi: 10.1136/emj.15.2.84. PMID 9570046
- [Background] Masel BE, DeWitt DS. Traumatic brain injury: a disease process, not an event. J Neurotrauma. 2010 Aug;27(8):1529-40. doi: 10.1089/neu.2010.1358. PMID 20504161
- [Background] Werner C, Engelhard K. Pathophysiology of traumatic brain injury. Br J Anaesth. 2007 Jul;99(1):4-9. doi: 10.1093/bja/aem131. PMID 17573392
- [Background] Carney N, Lujan S, Dikmen S, Temkin N, Petroni G, Pridgeon J, Barber J, Machamer J, Cherner M, Chaddock K, Hendrix T, Rondina C, Videtta W, Celix JM, Chesnut R. Intracranial pressure monitoring in severe traumatic brain injury in latin america: process and methods for a multi-center randomized controlled trial. J Neurotrauma. 2012 Jul 20;29(11):2022-9. doi: 10.1089/neu.2011.2019. Epub 2012 May 15. PMID 22435793
- [Background] Timofeev I, Carpenter KL, Nortje J, Al-Rawi PG, O'Connell MT, Czosnyka M, Smielewski P, Pickard JD, Menon DK, Kirkpatrick PJ, Gupta AK, Hutchinson PJ. Cerebral extracellular chemistry and outcome following traumatic brain injury: a microdialysis study of 223 patients. Brain. 2011 Feb;134(Pt 2):484-94. doi: 10.1093/brain/awq353. Epub 2011 Jan 18. PMID 21247930
- [Background] Sarrafzadeh AS, Sakowitz OW, Callsen TA, Lanksch WR, Unterberg AW. Bedside microdialysis for early detection of cerebral hypoxia in traumatic brain injury. Neurosurg Focus. 2000 Nov 15;9(5):e2. doi: 10.3171/foc.2000.9.5.2. PMID 16821754
- [Background] Nortje J, Gupta AK. The role of tissue oxygen monitoring in patients with acute brain injury. Br J Anaesth. 2006 Jul;97(1):95-106. doi: 10.1093/bja/ael137. Epub 2006 Jun 3. PMID 16751641
- [Background] Smielewski P, Coles JP, Fryer TD, Minhas PS, Menon DK, Pickard JD. Integrated image analysis solutions for PET datasets in damaged brain. J Clin Monit Comput. 2002 Dec;17(7-8):427-40. doi: 10.1023/a:1026293611455. PMID 14650638
- [Background] Vespa PM, McArthur D, O'Phelan K, Glenn T, Etchepare M, Kelly D, Bergsneider M, Martin NA, Hovda DA. Persistently low extracellular glucose correlates with poor outcome 6 months after human traumatic brain injury despite a lack of increased lactate: a microdialysis study. J Cereb Blood Flow Metab. 2003 Jul;23(7):865-77. doi: 10.1097/01.WCB.0000076701.45782.EF. PMID 12843790
- [Background] Verweij BH, Muizelaar JP, Vinas FC, Peterson PL, Xiong Y, Lee CP. Impaired cerebral mitochondrial function after traumatic brain injury in humans. J Neurosurg. 2000 Nov;93(5):815-20. doi: 10.3171/jns.2000.93.5.0815. PMID 11059663
- [Background] Nordstrom CH, Nielsen TH, Schalen W, Reinstrup P, Ungerstedt U. Biochemical indications of cerebral ischaemia and mitochondrial dysfunction in severe brain trauma analysed with regard to type of lesion. Acta Neurochir (Wien). 2016 Jul;158(7):1231-40. doi: 10.1007/s00701-016-2835-z. Epub 2016 May 17. PMID 27188288
- [Background] Lazaridis C, Robertson CS. The Role of Multimodal Invasive Monitoring in Acute Traumatic Brain Injury. Neurosurg Clin N Am. 2016 Oct;27(4):509-17. doi: 10.1016/j.nec.2016.05.010. PMID 27637400
- [Background] Faul M, Wald MM, Rutland-Brown W, Sullivent EE, Sattin RW. Using a cost-benefit analysis to estimate outcomes of a clinical treatment guideline: testing theBrain Trauma Foundation guidelines for the treatment of severe traumatic brain injury. J Trauma. 2007 Dec;63(6):1271-8. doi: 10.1097/TA.0b013e3181493080. PMID 18212649
- [Background] Hutchinson PJ, Jalloh I, Helmy A, Carpenter KL, Rostami E, Bellander BM, Boutelle MG, Chen JW, Claassen J, Dahyot-Fizelier C, Enblad P, Gallagher CN, Helbok R, Hillered L, Le Roux PD, Magnoni S, Mangat HS, Menon DK, Nordstrom CH, O'Phelan KH, Oddo M, Perez Barcena J, Robertson C, Ronne-Engstrom E, Sahuquillo J, Smith M, Stocchetti N, Belli A, Carpenter TA, Coles JP, Czosnyka M, Dizdar N, Goodman JC, Gupta AK, Nielsen TH, Marklund N, Montcriol A, O'Connell MT, Poca MA, Sarrafzadeh A, Shannon RJ, Skjoth-Rasmussen J, Smielewski P, Stover JF, Timofeev I, Vespa P, Zavala E, Ungerstedt U. Consensus statement from the 2014 International Microdialysis Forum. Intensive Care Med. 2015 Sep;41(9):1517-28. doi: 10.1007/s00134-015-3930-y. PMID 26194024
- See also: Head injury statistics in the UK — https://www.headway.org.uk/about-brain-injury/further-information/statistics/

DOCUMENTS (1):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT02993549/Prot_000.pdf